CLINICAL TRIAL: NCT02370654
Title: Chen-style Tai Chi in Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Saey, Didier, M.D. (Individual); Maltais, Francois, M.D. (Industry)
Responsible Party: Principal Investigator, Louis Gendron, MSc, Laval University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: TCCOPD CER21009
Record Dates: First submitted 2015-02-11; First posted 2015-02-25 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Tai chi; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi (Experimental): 12 week Tai chi intervention, 3 sessions per week, 90 minutes per session
  Interventions: Behavioral: Tai chi
- Conventional exercise (Active Comparator): 12 week conventional exercise intervention, 3 sessions per week, 90 minutes per session
  Interventions: Behavioral: Conventional exercise

INTERVENTIONS:
Behavioral: Tai chi
  Arms: Tai Chi
Behavioral: Conventional exercise
  Arms: Conventional exercise

SUMMARY:
This study will evaluate the effects of Chen-style Tai Chi compared to conventional exercise in pulmonary rehabilitation for COPD patients. Half of participants will receive the Chen-style Tai Chi intervention, while the other half will receive the conventional exercise intervention. Both groups will receive the same eduction and support during pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 between 30 and 80% of the predicted normal values
* FEV1/FVC ratio < 70%

Exclusion Criteria:

* Patients with very severe COPD (GOLD IV);
* Patients that had a COPD exacerbations within the preceding 2 weeks of the baseline assessments;
* Significant hypoxemia at rest or during exercise (SpO2 <85%);
* Already following a rehabilitation program;
* Have physical limitations that compromises participation to a Tai chi and a conventional exercise program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-03; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline dyspnea at 12 weeks | Baseline, 12 weeks
  Dyspnea will be assessed using the chronic respiratory questionnaire (CRQ)

SECONDARY OUTCOMES:
Change from baseline lung function at week 12 (Spirometry and whole-body plethysmography) | Baseline, 12 weeks
  Spirometry and whole-body plethysmography will be used for baseline and post-training (12 weeks) lung function testing.
Change from baseline walking distance at 12 weeks (distance walked during the six-minute walk test) | Baseline, 12 weeks
  The distance walked during the six-minute walk test will be used to evaluate the functional exercise capacity of all participants at baseline and post-rehabilitation.
Change from baseline exercise capacity at 12 weeks(Endurance time during a constant work rate bicycle ergometry exercise test) | Baseline, 12 weeks
  Endurance time during a constant work rate bicycle ergometry exercise test will be used to evaluate the exercise capacity of all participants at baseline and post-rehabilitation.
Change from baseline isokinetic quadriceps muscle function at 12 weeks | Baseline, 12 weeks
  Voluntary isokinetic quadriceps muscle function will be determined by quantification of force, endurance, and fatigability of the dominant quadriceps during a series of 30 repetitions at an angular velocity of 90°/s of a knee extension test.
Change from baseline isometric quadriceps muscle strength at 12 weeks (force of the dominant quadriceps will be measured during a single magnetic stimulation of the femoral nerve) | Baseline, 12 weeks
  The force of the dominant quadriceps will be measured during a single magnetic stimulation of the femoral nerve (Twitch force of the quadriceps [Twq]) and during a maximum voluntary contraction (MVC).
Change from baseline physical activity at 12 weeks (participants will be equipped with a physical activity monitor) | Baseline, 12 weeks
  To monitor physical activity, participants will be equipped with a physical activity monitor. The device will monitor the daily energy expenditure, the duration of physical activities above the pre-determined intensity level (Metabolic Equivalent of Task (MET) >3), and also the total daily number of steps.
Change from baseline quality of life (QoL) at 12 weeks | Baseline, 12 weeks
  In addition to dyspnea (primary outcome), the CRQ will be used also to measure other physical-functional limitations due to COPD with questions related to fatigue and energy levels.
Change from baseline health status at 12 weeks (determined with the COPD Assessment test (CAT). | Baseline, 12 weeks
  Impact of COPD on a person's life will be determined with the COPD Assessment test (CAT).
Change from baseline balance (Berg Balance Test (BBT) at 12 weeks | Baseline, 12 weeks
  The Berg Balance Test (BBT) will be used to evaluate the effect of the interventions on patient's balance.
Change from baseline of composite serum and plasma biomarkers at 12 weeks | Baseline, 12 weeks
  During the baseline assessment and after the rehabilitation program, blood samples from patients will be taken in order to investigate the effect of the interventions on different biomarkers related to systemic inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, PhD, Principal Investigator — Francois.Maltais@fmed.ulaval.ca
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada